CLINICAL TRIAL: NCT00821821
Title: A Phase IIa, Multi-centre, Randomised, Double-blind, Placebo Controlled, Clinical Study Investigating the Safety, Tolerability and Pharmacokinetics of MCI-186 in Subjects With Acute Ischemic Stroke
Brief Title: Safety and Pharmacokinetics of MCI-186 in Subjects With Acute Ischemic Stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MCI-186-E04
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Acute Ischemic Stroke (AIS)
MeSH Terms: conditions — Ischemic Stroke | interventions — Edaravone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MCI-186 (Experimental)
  Interventions: Drug: MCI-186
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MCI-186 — Cohort 1: Edaravone: circa 1000 mg / 72-hour infusion
  Cohort 2: Edaravone: circa 2000 mg / 72-hour infusion
  Other Names: Edaravone
  Arms: MCI-186
Drug: Placebo — Cohort1:circa 1000mg / 72-hour infusion matching placebo
  Cohort2:circa 2000mg / 72-hour infusion matching placebo
  Arms: Placebo Group

SUMMARY:
The objectives of this study are to assess the safety, tolerability and local tolerance, and to investigate the plasma levels and terminal elimination half life of MCI-186, and to review the routine clinical and neurological assessments data of MCI-186 in subjects with acute ischemic stroke.

ELIGIBILITY:
Inclusion Criteria:

* Full functional independence prior to the present stroke (as evidenced by a pre-morbid modified Rankin Scale score of 0-2
* Clinical diagnosis of acute stroke with CT scan ruling out intracranial hemorrhage
* Onset of symptoms within 1-24 hours of commencement of infusion of study drug
* Measurable deficit on NIHSS (as evidenced by a score of 3-15)
* Full consciousness (i.e. the score for NIHSS item 1a=0)
* Written valid informed consent is obtained from the subject or his/her next of kin or legal representative if the subject is fully conscious (i.e. the score for NIHSS item 1a = 0) but unable to read and/or sign the ICF, in accordance with National legislation and local IRB requirements

Exclusion Criteria:

* Subjects who are unlikely to complete the infusion of investigational product and/or are unlikely to undergo active medical management during that period due to a severe clinical condition
* Subjects with severe illness with life expectancy less than 6 months
* Body weight in excess of 120 kg
* Subjects who have received rTPA or other thrombolytics (e.g. urokinase, streptokinase, reteplase, tenecteplase) within the previous 24 hours
* Likelihood of forbidden concomitant therapy such as vascular surgery, coronary artery bypass graft (CABG), valve replacement, or carotid endarterectomy (CEA)
* Evidence of cerebral herniation
* Subjects with confounding neurological diseases such as dementia
* Subjects with CADASIL, Moya Moya, or carotid dissection
* Subjects who have experienced a stroke within the previous 3 months (Note: subjects who have recently experienced a TIA, but whose premorbid mRS prior to their stroke is 0-2, will be allowed to enter the study)
* Evidence from admission imaging tests of infarction involving >1/3 of MCA territory, or entire ACA territory involvement, or internal carotid artery (ICA) occlusions without coexisting separate occlusion of the middle cerebral artery (because of the difficulty distinguishing between chronic and acute ICA lesions in such subjects)
* Pathology other than cerebral infarction on any admission imaging tests (e.g. ICH or SAH, AV malformation, cerebral aneurysm, or cerebral neoplasm)
* Current or previous known excessive alcohol use or dependence
* Current known illicit drug use or dependence
* Participation in a previous clinical study within 30 days
* Subjects unlikely to be able and willing to attend all study follow-up visits
* Any other conditions which in the opinion of the investigator deem the subject ineligible for inclusion
* Females who are pregnant or intend to become pregnant or subjects (male and female) who do not agree to use effective contraception for 3 months after end of treatment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Study Chair — Information at Mitsubishi Pharma Europe
Locations (3):
- Helsinki University Central Hospital, Helsinki, Finland
- Erasmus Medical Center, Rotterdam, Netherlands
- Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle, United Kingdom

REFERENCES:
- [Result] Kaste M, Murayama S, Ford GA, Dippel DW, Walters MR, Tatlisumak T; MCI-186 study group. Safety, tolerability and pharmacokinetics of MCI-186 in patients with acute ischemic stroke: new formulation and dosing regimen. Cerebrovasc Dis. 2013;36(3):196-204. doi: 10.1159/000353680. Epub 2013 Oct 12. PMID 24135530

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-186 Cohort1: Edaravone: circa 1000 mg / 72-hour infusion
- MCI-186 Cohort2: Edaravone: circa 2000 mg / 72-hour infusion
- Placebo Group: Cohort1:circa 1000mg / 72-hour infusion matching placebo
  Cohort2:circa 2000mg / 72-hour infusion matching placebo
Period: Overall Study
Arm/Group | MCI-186 Cohort1 | MCI-186 Cohort2 | Placebo Group
Started | 12 | 13 | 11
Completed | 12 | 13 | 11
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MCI-186 Cohort1 | MCI-186 Cohort2 | Placebo Group | Total
Number analyzed (Participants) | 12 | 13 | 11 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 5 | 9 | 2 | 16
  >=65 years | 7 | 4 | 9 | 20
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 3 | 9
  Male | 10 | 9 | 8 | 27

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Experienced Adverse Events
Description: Additional Outcome Measures are included in Tables for Serious Adverse Events and Other Adverse Events to report their numbers and frequency.
Time Frame: 87days
Measure: Number; unit: participants
Arm/Group | MCI-186 Cohort1 | MCI-186 Cohort2 | Placebo Group
Number analyzed (Participants) | 12 | 13 | 11
participants
  Deaths | 0 | 0 | 0
  Serious Adverse Events | 0 | 2 | 1
  Other Adverse Events | 12 | 10 | 10

2. Secondary Outcome: Plasma MCI-186 Pharmacokinetics
Description: The geometric mean values of MCI-186 plasma concentration at the end of the infusion (at 72h) in cohorts 1 and 2 were determined.
Time Frame: 72 hours
Population: The subjects with reliable measured values for plasma concentration were selected for pharmacokinetic analysis: 5 subjects in MCI-186 Cohort 1 and 11 subjects in MCI-186 Cohort 2.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng / ml
Groups:
- MCI-186 Cohort1: Edaravone:circa 1000mg / 72-hour infusion
- MCI-186 Cohort2: Edaravone:circa 2000mg / 72-hour infusion
Arm/Group | MCI-186 Cohort1 | MCI-186 Cohort2
Number analyzed (Participants) | 5 | 11
ng / ml | 391 (24.21) [45.81 to 3338] | 1595 (51.57) [958.3 to 2655]

3. Secondary Outcome: mRS, NIHSS, Barthel Index
Time Frame: throughout study
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 87 days
Groups:
- MCI-186 Cohort1: Edaravone: circa 1000mg / 72-hour infusion
- MCI-186 Cohort2: Edaravone: circa 2000mg / 72-hour infusion
Arm/Group | MCI-186 Cohort1 | MCI-186 Cohort2 | Placebo Group
Serious Adverse Events (participants affected / at risk) | 0/12 | 2/13 | 1/11
Other Adverse Events (participants affected / at risk) | 12/12 | 10/13 | 10/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 Cohort1 (N=12) | MCI-186 Cohort2 (N=13) | Placebo Group (N=11)
Gout (Metabolism and nutrition disorders) | 0 | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-186 Cohort1 (N=12) | MCI-186 Cohort2 (N=13) | Placebo Group (N=11)
Atrial Fibrillation (Cardiac disorders) | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cataract (Eye disorders) | 0 | 0 | 1
Vision Blurred (Eye disorders) | 0 | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 5 | 1 | 2
Vomiting (Gastrointestinal disorders) | 1 | 0 | 1
Fatigue (General disorders) | 1 | 0 | 0
Infusion Site Phlebitis (General disorders) | 1 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Vessel Puncture Site Haematoma (General disorders) | 1 | 0 | 1
Eczema Infected (Infections and infestations) | 0 | 1 | 0
Groin Abscess (Infections and infestations) | 0 | 0 | 1
Infusion Site Infection (Infections and infestations) | 0 | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 1 | 0 | 0
Urinary Tract Infection (Infections and infestations) | 1 | 0 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 1 | 0
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 1
Blood Glucose Increased (Investigations) | 0 | 0 | 1
Blood Uric Acid Increased (Investigations) | 0 | 0 | 1
C-Reactive Protein Increased (Investigations) | 1 | 0 | 0
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 0 | 1
Hepatic Enzyme Increased (Investigations) | 1 | 0 | 0
Liver Function Test Abnormal (Investigations) | 0 | 0 | 1
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 | 1 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Cerebrovascular Accident (Nervous system disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1 | 0
Headache (Nervous system disorders) | 4 | 4 | 4
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Neuralgia (Nervous system disorders) | 1 | 1 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Simple Partial Seizures (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 0 | 0 | 1
Speech Disorder (Nervous system disorders) | 0 | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Urethral Haemorrhage (Renal and urinary disorders) | 0 | 0 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural Fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Stasis Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 3 | 2 | 4
Hypotension (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other